CLINICAL TRIAL: NCT02406235
Title: Evaluating a Novel Onco-genetic BRCA Testing Counselling Model Among Patients With Ovarian Cancer - ENGAGE Study
Brief Title: Evaluating a Novel Onco-genetic BRCA Testing Counselling Model Among Patients With Ovarian Cancer
Acronym: ENGAGE
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Collaborators: Optum, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: D0816R00006
Record Dates: First submitted 2015-03-23; First posted 2015-04-02 (Estimated); Last update posted 2017-09-19 (Actual); Status verified 2017-09

CONDITIONS: Epithelial Ovarian/Fallopian Tube/Primary Peritoneal Cancer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The overall objective of this study is to assess turnaround time, pre-BRCA test onco-genetic counselling quality and satisfaction with a new onco-genetic BRCA testing model.

DETAILED DESCRIPTION:
This will be a prospective observational study of patients diagnosed with epithelial ovarian/fallopian tube/primary peritoneal cancer prior to, or at enrolment in this study. The study is descriptive in nature and does not attempt to test any specific a priori hypotheses.

Clinical teams (physicians and nurses) will be trained to discuss BRCA testing with ovarian cancer patients who meet study criteria and consent to participate in the study. Patients will be recruited from participating sites in North America and Europe. Patients selected per the study inclusion and exclusion criteria will be consented for participation in the study. Patients will be recruited during an estimated 12 month period and participating patients will be followed from enrollment in the study until provision of BRCA test results, final genetics counselling, and completion of satisfaction survey or death. A case report form will be developed to collect information on the primary variable of interest (i.e., turnaround time), patient and disease characteristics, medical history, treatment patterns and outcome of the BRCA test. In addition, a survey will be developed to evaluate patient's assessment of pre- BRCA onco-genetic counseling quality and satisfaction with onco-genetic testing process.

Finally, surveys will be developed to evaluate oncologist (or oncology nurse) and genetic counselor's assessment of the processes associated with the onco-genetic testing pathway.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with epithelial ovarian/fallopian tube/primary peritoneal cancer
* Patients aged 18 years or older at ovarian cancer diagnosis
* Provision of written informed consent
* Patient is able to read, write, and understand the material presented to them as part of this study, per the discretion of the physician

Exclusion Criteria:

* Patients with low grade epithelial ovarian cancer or non-epithelial ovarian cancer
* Patients enrolled in an interventional clinical trial for ovarian cancer or other malignancy at the time of conduct of this study
* Patients with BRCA testing any time prior to the study enrollment

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients diagnosed with epithelial ovarian/fallopian tube/primary peritoneal cancer prior to, or at enrolment in this study
Sampling Method: Probability Sample
Enrollment: 710 (Actual)
Dates: Start 2015-04-21 (Actual); Primary Completion 2016-09-30 (Actual); Study Completion 2016-09-30 (Actual)

PRIMARY OUTCOMES:
Assessing turnaround time with the new BRCA-testing pathway | participating patients will be followed from enrollment in the study until provision of BRCA test results, final genetics counselling and completion of satisfaction survey or death, an expected average of 2 months
  The primary objectives include a) assessing turnaround time with the new BRCA (Breast Cancer)-testing pathway; b) patient's assessment of pre-BRCA test onco-genetic counselling quality and satisfaction with the onco-genetic BRCA testing pathway; c) oncologists, and genetic counsellor's assessment of onco-genetic BRCA testing process. The study will be limited to patients with a diagnosis of ovarian cancer.

CONTACTS AND LOCATIONS:
Locations (26):
- United States (11):
  - Research Site, San Francisco, California
  - Research Site, Gainesville, Florida
  - Research Site, Sarasota, Florida
  - Research Site, Augusta, Georgia
  - Research Site, Worcester, Massachusetts
  - Research Site, Hackensack, New York
  - Research Site, Lake Success, New York
  - Research Site, Mineola, New York
  - Research Site, The Bronx, New York
  - Research Site, Chapel Hill, North Carolina
  - Research Site, Providence, Rhode Island
- Italy (7):
  - Research Site, Brescia, IT
  - Research Site, Genova, IT
  - Research Site, Milan, IT
  - Research Site, Modena, IT
  - Research Site, Napoli, IT
  - Research Site, Roma, IT
  - Research Site, Torino, IT
- Spain (8):
  - Research Site, A Coruña, SP
  - Research Site, Barcelona, SP
  - Research Site, Cáceres, SP
  - Research Site, Córdoba, SP
  - Research Site, Madrid, SP
  - Research Site, Murcia, SP
  - Research Site, Palma de Mallorca, SP
  - Research Site, Zaragoza, SP

REFERENCES:
- [Derived] Colombo N, Huang G, Scambia G, Chalas E, Pignata S, Fiorica J, Van Le L, Ghamande S, Gonzalez-Santiago S, Bover I, Grana Suarez B, Green A, Huot-Marchand P, Bourhis Y, Karve S, Blakeley C. Evaluation of a Streamlined Oncologist-Led BRCA Mutation Testing and Counseling Model for Patients With Ovarian Cancer. J Clin Oncol. 2018 May 1;36(13):1300-1307. doi: 10.1200/JCO.2017.76.2781. Epub 2018 Mar 20. PMID 29558274
- See also: D0816R00006_CSR_Synopsis.pdf — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=3060&filename=D0816R00006_CSR_Synopsis.pdf